CLINICAL TRIAL: NCT06217289
Title: Multicentric Study on Knowledgement and Behaviors of Health Care Professionals Handling Oral Solid Pharmaceutical Forms/Drugs
Brief Title: A Study on Behavior of Healthcare Professionals Who Handle Oral Solid Drug
Status: Completed | Type: Observational
Sponsor: Enrico Tomasi (Other)
Responsible Party: Sponsor-Investigator, Enrico Tomasi, Doctor, IRCCS San Raffaele
Organization: IRCCS San Raffaele (Other)
Other Study IDs: Recommendation n°19
Record Dates: First submitted 2024-01-02; First posted 2024-01-22 (Actual); Last update posted 2024-01-22 (Actual); Status verified 2024-01

CONDITIONS: Behavior
MeSH Terms: conditions — Behavior | interventions — Observation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Observation — Observation and knowledgement on behavior of healthcare professional workers during hpreparation of oral solid pharmaceutical drug

SUMMARY:
A study on behavior of healthcare professionals who handle oral solid drug

DETAILED DESCRIPTION:
A study on behavior of healthcare professionals who handle oral solid drug

ELIGIBILITY:
Inclusion Criteria:

• Healthcare professionals in charge of drug preparation

Exclusion Criteria:

• There are not exclusion criteria

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Healthcare professionals in charge of drug preparation
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2021-09-15 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Observation on behavior of healthcare professional workers during hpreparation of oral solid pharmaceutical drug | 3 months
  Observation on behavior of healthcare professional workers during hpreparation of oral solid pharmaceutical drug

CONTACTS AND LOCATIONS:
Overall Officials: Maria Fazio, Principal Investigator — IRCCS
Locations (1):
- IRCCS Ospedale San Raffaele, Milan, Italy

IPD SHARING:
Plan to Share IPD: No